CLINICAL TRIAL: NCT02928679
Title: Multi-parametric Imaging of the Knee in Obese Patients With Knee Osteoarthritis Following Liraglutide Treatment, Investigating the Impact on Inflammation
Brief Title: Multi-parametric Imaging of the Knee in Obese Patients With Knee Osteoarthritis; Weight Maintenance
Acronym: IM-LOSEIT-II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henrik Gudbergsen (Other)
Responsible Party: Sponsor-Investigator, Henrik Gudbergsen, MD, PhD, Parker Research Institute
Organization: Parker Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 137.05
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis; Obesity
Keywords: Magnetic resonance imaging; Dynamic contrast enhanced MRI; Liraglutide 3 mg; Liraglutide; Obesity; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Obesity | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide 3 mg (Experimental): Arm description: Subjects will be up titrated to liraglutide 3 mg QD and stay on that dose for the remainder of the 52-week drug intervention period.
  Drug: Liraglutide 3 mg QD administered in a 6 mg/mL, 3 mL pen for subcutaneous injection.
  Dose escalation scheme: Initial dosage of 0.6 mg per day, escalated bi-weekly by 0.6 mg to 3 mg per day over a total of 8 weeks.
  Interventions: Drug: Liraglutide 3 mg (Saxenda)
- Liraglutide 3 mg placebo (Placebo Comparator): Arm description: Subjects will be up titrated to liraglutide 3 mg placebo QD and stay on that dose for the remainder of the 52-week drug intervention period.
  Drug: Liraglutide 3 mg placebo QD administered in a 6 mg/mL drug equivalent volumes, 3 mL pen for subcutaneous injection.
  Dose escalation scheme: Initial dosage of a 0.6 mg drug equivalent volume per day, escalated bi-weekly by an 0.6 mg drug equivalent volume per day to a 3 mg drug equivalent volume per day over a total of 8 weeks.
  Interventions: Drug: Liraglutide 3 mg placebo

INTERVENTIONS:
Drug: Liraglutide 3 mg (Saxenda)
  Arms: Liraglutide 3 mg
Drug: Liraglutide 3 mg placebo
  Arms: Liraglutide 3 mg placebo

SUMMARY:
This is a substudy to a randomised trial investigating the effect of liraglutide on body weight and pain in overweight or obese patients with knee osteoarthritis (NCT02905864). In the parent trial, patients will be subjected to an 8-week diet intervention phase including a low-calorie diet and dietetic counseling, after which patients will be randomised to receive either liraglutide 3 mg or liraglutide 3 mg placebo as an add-on to dietetic guidance on re-introducing regular foods and a focus on continued motivation to engage in a healthy lifestyle.

This substudy aims to investigate the impact of, and subsequent change of, joint inflammation, articular cartilage composition, overall knee morphology, and clinical symptoms, in obese patients with knee osteoarthritis following a randomisation to Liraglutide 3 mg or Liraglutide 3 mg placebo treatment between weeks 0-52.

ELIGIBILITY:
Inclusion Criteria:

* Same as parent trial (NCT02905864)

Further Exclusion Criteria:

* Same as parent trial (NCT02905864)
* Usual exclusion criteria for MRI (i.e. pacemakers etc.)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-02-20 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Change in the degree of inflammation in the knee-joint (DCE-MRI) | Week 0 to 52
  Change will be assessed via a dynamic contrast enhanced MRI evaluation of corpus hoffa (Ballegaard C et al. and Riis RG et al.)

SECONDARY OUTCOMES:
Change in the degree of inflammation in the knee-joint (CE-MRI) | Week 0 to 52
  Change will be assessed via a static contrast enhanced MRI evaluation of the level of synovitis in the knee-joint (11 sites scored 0-2, ad modum Guermazi et al.)
Change in the degree of inflammation in the knee-joint (MRI) | Week 0 to 52
  Change will be assessed via a conventional MRI evaluation of the level of synovitis and effusion (combined) in the knee-joint (MOAKS)
Change in cartilage composition | Week 0 to 52
  Change will be assessed via T2-maps of cartilage in the weight-bearing parts of the knee-joint (ROI)
Change in bone marrow lesions | Week 0 to 52
  Change will be assessed via the MRI knee scoring system MOAKS; BML sum-score

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute and Department of Radiology at Bispebjerg and Frederiksberg Hospital, Frederiksberg, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No